CLINICAL TRIAL: NCT01775540
Title: Study to Evaluate the Ocular Surface Healing Action of the Artificial Tear Systane ULTRA Using Both Positive (Maxidex) and Negative (Saline Solution) Controls
Brief Title: Systane Ultra Versus Maxidex Versus Saline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Penny Asbell, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 11-1230
Record Dates: First submitted 2012-12-07; First posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Dry Eye Disease
Keywords: Dry eye; Artificial tears; Ocular surface inflammation
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops; Saline Solution; Dexamethasone; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Systane Ultra (Experimental): Artificial tear Eyedrop, 1 drop used four times a day (QID) for 4 weeks
  Interventions: Drug: Systane Ultra
- Saline solution (Placebo Comparator): Saline solution Eyedrop, 1 drop used QID for 4 weeks
  Interventions: Drug: Saline solution
- Maxidex (Active Comparator): Steroid eyedrop, 1 drop QID for 4 weeks
  Interventions: Drug: Maxidex

INTERVENTIONS:
Drug: Systane Ultra — Artificial tear Eyedrop, 1 drop used QID for 4 weeks
  Other Names: Artificial Tears
  Arms: Systane Ultra
Drug: Saline solution — Saline solution,1 drop used QID for 4 weeks
  Arms: Saline solution
Drug: Maxidex — Eyedrop-1 drop QID for 4 weeks
  Other Names: Dexamethasone 0.1% eyedrop
  Arms: Maxidex

SUMMARY:
This study was to evaluate the healing action on the eye surface of the artificial tear Systane® ULTRA as compared to two other eyedrops: Maxidex and Saline solution. Dry eye disease leads to inflammation of the eye surface and treating dry eyes with artificial tears may lead to reduction in this inflammation and improvement of symptoms and signs.

DETAILED DESCRIPTION:
For all patients who present to the office with a history of dry eyes:

1. Consent forms will be obtained from every patient. Informed consent will be discussed with the patient in detail. Every topic will be addressed separately. All risks, benefits, and alternatives will be discussed. Patient will be allowed to ask questions, and all questions will be answered. The assessment will be made after that conversation, whether or not the patient understood the consent as described above. Each subject will be allowed as much time as needed to review and sign the consent forms.
2. All patients will be asked to fill out the Ocular Surface Discomfort Index (OSDI) questionnaire to ensure they meet the inclusion criteria. If patients score meets eligibility requirements a general and ocular history will be taken. (Time: 10 min)
3. A pregnancy test will be given to all female subjects of child bearing age. A standard eye exam will be performed to rule out any other ocular pathology besides refractive error. This allows for confirmation that all study subjects have dry eye disease. Topical fluorescein and lissamine dye will be used to record staining on the cornea and conjunctiva of subjects as well as the tear film break-up time (TFBUT). Both of these dyes are used as standard-of-care in eye exams around the country. TFBUT will first be determined through application of sodium fluorescein onto the eye using DET strip. Following triplicate evaluation of TFBUT in each eye, ocular staining will be determined with liquid fluorescein and lissamine dyes administered in liquid form. (Time 15 min).
4. Patients will be given Alcon questionnaires to fill out, inquiring about past treatments, daily symptoms and distress associated with their dry eye disease. (Time:15 minutes) This also serves as a waiting period for some of the dye to wash out.
5. Using a graduated disposable 5 µl microcapillary tube (Wiretol-Micropipettes, Drummond Scientific Co., Broomall, PA, USA) up to 5 µl of tears / eye will be collected from the inferior temporal tear meniscus of each participant, without corneal anesthesia, taking care to ensure that the lid margin and corneal surface were not touched. A maximum of 5 minutes will be allowed per eye for collection of minimal 5 uL of tear. Tears will be immediately dispensed into pre-labeled Eppendorf tubes and placed on dry ice until transferred to -80oC for storage. (Time: 10 minutes)
6. A technique known as Impression Cytology (IC) will be used to isolate epithelial cells from the conjunctiva. Anesthetic drops will be administered to each eye before the procedure. Blunted forceps are used to gently press a piece of filter paper against the patient's conjunctiva. The paper is gently lifted off, and sent to the Mount Sinai Laboratory for analyses. (Estimated collection time: 15 minutes). A total of 6 pieces per patient (3 pieces per eye) will be collected on each scheduled visit. For HLA-DR analysis, 2 pieces from each eye will be held at room temperature in a vial containing fixative until assay. The remaining 1 piece from each eye will be pooled together in one vial for RT-PCR assays in the following order: (1) immediately merged into a pre-labeled Eppendorf tube with 600 µL of TriZol Reagent; (2) Vortex for 30 seconds; (3) sealed with Saran Wrap; (4) transfer to -80C for storage until assay.
7. Measurement of Intraocular pressure using Tonopen.
8. As a part of the substudy we intend to treat patients with Systane ULTRA®, Maxidex, (both of which are FDA approved ophthalmic solutions), or the saline solution placebo. Subjects will be assigned to one of the three groups as per randomization sequence and the corresponding eye drop will be dispensed.
9. The patient's response to treatment will be assessed after approximately 4 weeks (+/- 5 days) using the same diagnostic tests in order to assess the sensitivity of these diagnostic tests to detect the response to medical treatment of dry eye disease. In addition to baseline and 4 week visits, safety evaluations will be performed at a 2 week (+/- 5 days) visit. All the procedures done during the baseline visit will be repeated except pregnancy test, tear collection and impression cytology.

ELIGIBILITY:
Inclusion Criteria:

* A score of at least 15 on the Ocular Surface Discomfort Index (OSDI) symptom questionnaire.
* Moderate vital staining, fluorescein (for corneal evaluation, 3-15 on the NEI scale) OR lissamine (for conjunctival evaluation, score of 2-6; temporal and nasal areas, each graded 0-3).
* Willingness to use study drugs 4 times per day in both eyes.
* Willingness to discontinue use of other artificial tear products.
* Patient must provide written informed consent
* Patient must understand the scope of the study including completion of worksheet and be willing to follow instructions and return for all required study visits
* An intraocular pressure less than or equal to 22 mmHg in both eyes

Exclusion Criteria:

* Contact Lens wearers
* Pregnant and/or lactating women
* Those with moderate to severe Meibomian Gland Disease i.e. plugging of 3 or more glands and/or pasty secretion from 3 or more glands or presence of obstructed glands out of a total of 10 glands evaluated in the central portion of the lower lid.
* Uncontrolled systemic or ocular disease
* Dry eye due to seasonal allergic conjunctivitis, contact lens related conjunctivitis or other acute or seasonal diagnosis.
* Are monocular and/or legally blind
* Had ocular surgery or trauma within last six months
* Participation in an ophthalmic drug or device research study within 30 days prior to entry in this study
* Current use of any eye drops other than artificial tears
* Use of Restasis within three months prior to entry in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
OSDI score | at Baseline
  questionnaire pertaining to dry eye symptoms answered by patients
OSDI score | visit 2 (at 2 weeks)
  questionnaire pertaining to dry eye symptoms answered by patients
OSDI score | at visit 3 (at 4 weeks)
  questionnaire pertaining to dry eye symptoms answered by patients

SECONDARY OUTCOMES:
Tear Film break up time | at Baseline
  Time taken for the first dry spot to appear in the tear film
Tear Film break up time | at visit 2 (at 2 weeks)
  Time taken for the first dry spot to appear in the tear film
Tear Film break up time | at visit 3 (at 4 weeks)
  Time taken for the first dry spot to appear in the tear film
Corneal Staining | at Baseline
  Grading of fluorescein staining of the cornea using a slit lamp and NEI grading scale
Corneal Staining | at visit 2 (at 2 weeks)
  Grading of fluorescein staining of the cornea using a slit lamp and NEI grading scale
Corneal Staining | at visit 3 (at 4 weeks)
  Grading of fluorescein staining of the cornea using a slit lamp and NEI grading scale
Conjunctival Staining | at Baseline
  Grading of Lissamine green staining of the conjunctiva using a slit lamp and NEI grading scale
Conjunctival Staining | at visit 2 (at 2 weeks)
  Grading of Lissamine green staining of the conjunctiva using a slit lamp and NEI grading scale
Conjunctival Staining | at visit 3 (at 4 weeks)
  Grading of Lissamine green staining of the conjunctiva using a slit lamp and NEI grading scale
Best corrected visual acuity | at Baseline
  BSCVA using ETDRS charts
Best corrected visual acuity | at visit 2 (at 2 weeks)
  BSCVA using ETDRS charts
Best corrected visual acuity | at visit 3 (at 4 weeks)
  BSCVA using ETDRS charts
Tear Cytokines | At baseline
  Tear samples collected from both eyes using microcapillary tube. Samples analysed for inflammatory cytokines using Luminex bioassays
Tear Cytokines | At visit 3 (at 4 weeks)
  Tear samples collected from both eyes using microcapillary tube. Samples analysed for inflammatory cytokines using Luminex bioassays
mRNA for HLA-DR | At baseline
  Cell samples collected via impression cytology and analysed for mRNA expression via flowcytometer
mRNA for HLA-DR | At visit 3 (at 4 weeks)
  Cell samples collected via impression cytology and analysed for mRNA expression via flowcytometer
HLA-DR expression | At baseline
  Cell samples collected via impression cytology and analysed for HLA-DR expression via flowcytometer
HLA-DR expression | At visit 3 (at 4 weeks)
  Cell samples collected via impression cytology and analysed for HLA-DR expression via flowcytometer
IDEEL questionnaire | At baseline
  questionnaire pertaining to dry eye symptoms, quality of life, and treatment answered by patients
IDEEL questionnaire | At visit 2 (at 2 weeks)
  questionnaire pertaining to dry eye symptoms, quality of life, and treatment answered by patients
IDEEL questionnaire | At visit 3 (at 4 weeks)
  questionnaire pertaining to dry eye symptoms, quality of life, and treatment answered by patients

CONTACTS AND LOCATIONS:
Overall Officials: Penny Asbell, MD, MBA, FACS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States